CLINICAL TRIAL: NCT02304510
Title: Prevalence of Heavy Menstrual Bleeding in Female Population Living in Beijing
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Siyan Zhan, Professor, Peking University
Other Study IDs: PEKU-BJ-2014
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Menorrhagia
Keywords: Prevalence; Menorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- females: females aged between 18 and 50 years old living in Beijing

SUMMARY:
The purpose of the study is to estimate the prevalence of heavy menstrual bleeding (HMB) in females aged between 18 and 50 years old living in Bejing.

DETAILED DESCRIPTION:
This study is an observational, cross-sectional study. A representative sample of 2800 eligible women with different occupations such as farmers, service providers, workers, professional specialists, students and civil servants will be recruited. A cluster sampling method with probability proportional to the distribution of occupation in women in Beijing will be used. Demographic data will be collected by questionnaire. Menstrual bleeding will be evaluated by Pictorial Blood loss Assessment Chart (PBAC). According to the international definition of HMB, a PBAC score more than 100 is considered as HMB.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 18 and 50 years (inclusive)
* Stay in Beijing for more than 6 months
* Signed ICF was obtained

Exclusion Criteria:

* Not achieve the menarche
* With the last menstruation more than one year ago
* Experienced amenorrhea, currently take hormone therapy to induce menstruation
* Had undergone a hysterectomy
* Currently breastfeeding a baby
* Being pregnant

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: residents of Beijing
Sampling Method: Probability Sample
Enrollment: 2455 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of HMB | from date of inclusion until the end of the study currently planned (about 7 months)

SECONDARY OUTCOMES:
Prevalence of HMB in different subgroups | from date of inclusion until the end of the study currently planned (about 7 months)
  Subgroups include groups with different age, occupations, education levels, fertility status, with/without combined gynecological diseases.
Identify risk factors associated with HMB | from date of inclusion until the end of the study currently planned (about 7 months)
  Identified HMB subjects will be assigned into the case group. Non-HMB subjects will be assigned into the control group. Logistic regression model will be carried out to analyze the associations between possible demographic factors and risk of HMB by calculating odds ratios (OR) with 95% confidence intervals (CIs).

CONTACTS AND LOCATIONS:
Overall Officials: Siyan Zhan, MD,PhD, Principal Investigator — Peking University Health Science Center
Locations (1):
- Peking University Health Science Center, Beijing, China